CLINICAL TRIAL: NCT01520350
Title: Low-Dose Adjunctive Aripiprazole in the Treatment of Bipolar Depression: Double-Blind Placebo-Controlled Pilot Study
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: recruitment issues
Sponsor: Serge Beaulieu (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Serge Beaulieu, Medical Chief, Bipolar Disorders Program, Douglas Mental Health University Institute
Organization: Douglas Mental Health University Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARI_1109
Record Dates: First submitted 2012-01-25; First posted 2012-01-27 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Bipolar Disorder; Depressive Episode
MeSH Terms: conditions — Bipolar Disorder | interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mood stabilizer + Aripiprazole (Experimental)
  Interventions: Drug: Low dose Adjunctive Aripiprazole
- Mood stabilizer + placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Low dose Adjunctive Aripiprazole — low-dose 2-5mg/d for 8 weeks
  Other Names: Abilify
  Arms: Mood stabilizer + Aripiprazole
Drug: placebo — Placebo
  Arms: Mood stabilizer + placebo

SUMMARY:
Aripiprazole is a new antipsychotic agent which possesses unique capabilities compared to other antipsychotic agents, especially because of its partial dopaminergic agonistic activity. Moreover, like the other atypical agents, aripiprazole is an antagonist of the 5-HT2a receptor, and an agonist of the 5-HT1a receptor. These pharmacological properties should enable this molecule to provide antidepressant potentiating capabilities based on what has been observed with other compounds sharing similar pharmacological profiles.

Aripiprazole is now well recognized for its capacity to potentiate antidepressants in the treatment of unipolar depression. However, two randomized controlled trials of aripiprazole in the treatment of bipolar depression were negative. This surprising result may stem from the fact that the doses of aripiprazole used in these studies were rather high (17.6 ± 8.3 mg/d in study 1 and 15.5 ± 7.5 mg/d in study 2) and could have contributed to inhibit dopaminergic activity in key brain areas involved in the modulation of rewards, motivation and concentration. Bipolar depression is indeed heavily loaded with general symptoms of psychomotor retardation including poor concentration, low energy level, hypersomnolence, and hyperphagia. All these functions are modulated by dopamine and strategies aimed at improving dopaminergic function are used frequently to resolve residual symptoms of bipolar depression.

It is expected that aripiprazole used at a more adequate lower dose than in previous studies, should be efficacious in the treatment of bipolar type I depression.

ELIGIBILITY:
Inclusion Criteria:

* Age : 18-65
* Male or female
* Bipolar Disorder type I
* Current depressive episode (with MADRS ≥ 20 and item 2 (reported sadness) ≥ 3) for a minimum of 2 weeks but ≤ 52 weeks at screening visit and baseline visit)
* If female and of childbearing potential, is using an adequate method of contraception.
* Is treated with a mood stabilizer (lithium and/or valproate)
* Patient is able to give his consent

Exclusion Criteria:

* Is at high risk of suicide as defined by a score of ≥ 3 to item 10 of MADRS and/or in the clinical opinion of the investigator
* Hypo(mania) episode with YMRS ≥ 8
* Psychotic symptoms as defined by a score of ≥ 4 to item 8 (content) of YMRS and/or in the opinion of the investigator
* Is treated with fluoxetine OR lamotrigine OR carbamazepine OR any antidepressants
* Is treated with risperidone OR olanzapine OR quetiapine OR ziprazidone OR any antipsychotics
* Is pregnant or lactating or absence of contraceptive treatment
* Drug abuse or dependence as per DSM-IV (MINI)
* Unstable medical condition
* Other psychiatric condition, organic brain disorder, unstable and/or untreated medical condition such as hypothyroidism, hyperthyroidism, diabetes, cardiac condition, hypertension
* Deficit in vitamin B12 or folate
* Alcohol or drug abuse
* Rapid cycling (more than 4 mood episodes per year)
* Active or history of difficulty to swallow
* Seizures not currently controlled with medications
* Orthostatic hypotension
* A history of clinically significant cardiovascular disorders and cardiac arrhythmias
* A low white blood cell count
* Known eye disease
* Involuntary, irregular muscle movements, especially in the face
* Known hypersensitivity to aripiprazole and any components of its formulation
* Known lactose intolerance or have hereditary galactose intolerance or glucose-galactose malabsorption, because ABILIFY tablets contain lactose

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Response rate | 8 weeks
  The primary outcome measure will be the response rate as defined by a differential reduction of 5 points on the Montgomery Asberg rating Scale (MADRS) between the active treatment group and the placebo group at 8 weeks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Serge Beaulieu, MD, PhD, Principal Investigator — Douglas Institute
Locations (1):
- Douglas Mental Health University Institute, Montreal, Quebec, Canada